CLINICAL TRIAL: NCT00707447
Title: Evaluation of a Teaching and Treatment Programme for Primary Prevention of Type 2 Diabetes
Brief Title: Evaluation of a Primary Type 2 Diabetes Prevention Programme
Acronym: PREDIAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Collaborators: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Norbert Hermanns, PhD, Forschungsinstitut der Diabetes Akademie Mergentheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIDAM 006-04
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes-prevention; lifestyle modification; behavior therapy; self-management
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1/Control (Placebo Comparator): Control group received written information about diabetes risks with instructions about healthy eating and increasing physical exercise
  Interventions: Behavioral: Control
- 2/PREDIAS (Experimental): Intervention consists of a group programme (PREDIAS) aiming at modification of lifestyle
  Interventions: Behavioral: PREDIAS

INTERVENTIONS:
Behavioral: PREDIAS — Group programme aiming at modification of lifestyle: lifestyle changes, 12 lesson a 90 minutes, delivered in a group setting, consists of analysis of barriers against lifestyle changes, behavior analysis of eating and exercise behavior, modification of unhealthy lifestyle and relapse prevention
  Arms: 2/PREDIAS
Behavioral: Control — Written Information about diabetes risks. Brochure about the value of a healthy lifestyle, calorie table, suggestions for healthy food and daily exercise
  Arms: 1/Control

SUMMARY:
A type 2 diabetes prevention programme, named PREDIAS was developed. It consists of 12 lessons delivered as group sessions. Die efficacy of PREDIAS was studied in a randomized controlled study with 12 month follow up. Control group received written information about diabetes risk. Primary outcome variable was weight reduction at 12 months follow up. Secondary variables were impact of the intervention on glycemic parameters, lipids, eating and exercise behavior and other metabolic risk factors

DETAILED DESCRIPTION:
The PREDIAS programme was developed based on the interventions used in the Diabetes Prevention Study (DPS, Finland) and the Diabetes Prevention Programme (DPP; USA). The main purpose of PREDIAS was to develop a prevention programme delivered as a group programme to improve cost-benefit ration of diabetes prevention programmes.

ELIGIBILITY:
Inclusion Criteria:

* impaired fasting glucose and/or
* impaired glucose tolerance
* overweight (BMI > 26 kg/m²)

Exclusion Criteria:

* type 2 diabetes
* severe illness (cancer diagnosis, stroke or myocardial infarction in the last 12 months)
* diagnosis of a current mental disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2004-04; Primary Completion 2005-12 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, PhD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim
Locations (1):
- Research Institute of the Diabetes Academy Mergentheim (FIDAM), Bad Mergentheim, Germany

REFERENCES:
- [Result] Kulzer B, Hermanns N, Gorges D, Schwarz P, Haak T. Prevention of diabetes self-management program (PREDIAS): effects on weight, metabolic risk factors, and behavioral outcomes. Diabetes Care. 2009 Jul;32(7):1143-6. doi: 10.2337/dc08-2141. Epub 2009 Jun 9. PMID 19509014

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/Control: Control group received written instruction about healthy eating and increasing physical exercise
Period: Overall Study
Arm/Group | 1/Control | 2/PREDIAS
Started | 89 | 93
Completed | 81 | 85
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/Control | 2/PREDIAS | Total
Number analyzed (Participants) | 89 | 93 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 80 | 152
  >=65 years | 17 | 13 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.7) | 56.6 (9.6) | 56.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 78
  Male | 49 | 55 | 104
Region of Enrollment [Number; unit: participants]
  Germany | 89 | 93 | 182

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Mean weight change (in kg) after 12 months
Time Frame: 12 month
Population: Intention to treat analysis (LOCF) and per protocol analysis for primary outcome and per protocol analysis for secondary outcome measures
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Lifestyle Intervention Group (PREDIAS): 10 group sessions about healthy eating, modifying eating behavior, increasing physical activity and modifying risk factors for diabetes
- Control Group: Written information material about diabetes prevention by loosing weight, increasing physical activity
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
kg | -3.8 (5.2) | -1.4 (4.0)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; independent t-tests for between group comparisons, dependent t-tests for within group comparisons; Test type: Superiority or Other; p < .05, t-test, 2 sided — There was only one primary outcome variable, thus no adjustments for multiple comparisons were made

2. Primary Outcome: Waist Circumference
Description: Mean change in waist circumference (in cm) after 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
cm | -4.1 (6.0) | -0.4 (6.2)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; independent t-tests for between group comparisons, dependent t-tests for within group comparisons; Test type: Superiority or Other; p < .05, t-test, 2 sided

3. Secondary Outcome: Fasting Glucose
Description: Mean changes in fasting glucose (in mg/dl) after 12 month
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
mg/dl | -4.3 (11.3) | 1.8 (13.1)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; Test type: Superiority or Other; p < .05, t-test, 2 sided

4. Secondary Outcome: Glucose Tolerance
Description: Mean change in 2 hour postprandial oral glucose tolerance test (oGTT) (in mg/dl) after 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
mg/dl | -7.3 (30.8) | -8.2 (36.9)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; Test type: Superiority or Other; p < .05, t-test, 2 sided

5. Secondary Outcome: Physical Exercise
Description: Mean changes in physical exercise (in min/week) after 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
minutes per week | 46.6 (95.5) | 17.9 (63.8)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; Test type: Superiority or Other; p < .05, t-test, 2 sided

6. Secondary Outcome: Eating Behavior (TFEQ) - Cognitive Restraint
Description: The Three-Factor Eating Questionnaire (TFEQ) is a questionnaire used to assess food intake-behavior related research. The three factors of the TFEQ are: dietary restraint, disinhibition and hunger. The TFEQ contains 51 dichotomous Items (apply/ doesn't apply). The subscale "cognitive restraint" consists of 21 Item with a minimum score of "0" and a maximum score of "21". Low scores indicate an uninhibited eating behavior.
  Mean change in the TFEQ - cognitive restraint scale after 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
units on a scale | 3.9 (3.8) | 1.5 (3.0)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; Test type: Superiority or Other; p < .05, t-test, 2 sided

7. Secondary Outcome: Eating Behavior (TFEQ) - Disinhibition
Description: The Three-Factor Eating Questionnaire (TFEQ) is a questionnaire used to assess food intake-behavior related research. The three factors of the TFEQ are: dietary restraint, disinhibition and hunger. The TFEQ contains 51 dichotomous Items (apply/ doesn't apply). The subscale "disinhibition" consists of 16 Item with a minimum score of "0" and a maximum score of "16". High scores indicate an uninhibited eating behavior strongly depending on external cues.
  Mean change in the TFEQ - disinhibition scale after 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
units on a scale | -1.2 (2.7) | -0.4 (2.6)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; Test type: Superiority or Other; p < .05, t-test, 2 sided

8. Secondary Outcome: Eating Behavior (TFEQ) - Hunger
Description: The Three-Factor Eating Questionnaire (TFEQ) is a questionnaire used to assess food intake-behavior related research. The three factors of the TFEQ are: dietary restraint, disinhibition and hunger. The TFEQ contains 51 dichotomous Items (apply/ doesn't apply). The subscale "hunger" consists of 14 Item with a minimum score of "0" and a maximum score of "14". Low scores indicate an eating behavior strongly depending on feelings of hunger.
  Mean change in the TFEQ - hunger scale after 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
units on a scale | -1.1 (3.1) | -0.2 (2.7)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; Test type: Superiority or Other; p < .05, t-test, 2 sided

9. Secondary Outcome: Psychological Well-being (WHO-5)
Description: The WHO (Five) Well-being index consists of 5 items on the overall well-being over the last two weeks. Each of the five items is rated from 0 (= not present) to 5 (= constantly present). Scores are summated, with raw score ranging from 0 to 25. Then the scores are transformed to 0-100 by multiplying by 4, with higher scores meaning better well-being.
  Mean change in psychological well-being score (WHO-5) after 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
units on a scale | 1.4 (3.9) | 0.0 (4.2)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; Test type: Superiority or Other; p < .05, t-test, 2 sided

10. Secondary Outcome: Emotional Well-being/ Depression (CES-D)
Description: The Center for Epidemiologic Studies Depression Scale (CES-D) consists of 20 items scored from "0" to "3". Scores are summated, with raw score ranging from 0 to 25. Higher Scores idicate a higher depressive state.
  Mean change in depression score (CES-D) after 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Intervention Group (PREDIAS) | Control Group
Number analyzed (Participants) | 85 | 81
units on a scale | -3.5 (7.1) | -1.0 (6.1)
Statistical Analysis 1: Comparison: Lifestyle Intervention Group (PREDIAS) vs Control Group; Test type: Superiority or Other; p < .05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Description: The occurence of (serious) adverse events was assessed at each visit and at study close-out visit after 12 months
Groups:
- 2/PREDIAS: Intervention consists of a group programme (PRAEDIAS) aiming at modification of lifestyle
Arm/Group | 1/Control | 2/PREDIAS
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/85
Other Adverse Events (participants affected / at risk) | 0/81 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes